CLINICAL TRIAL: NCT03287661
Title: A Randomized Controlled Trial of an Online Chronic Pain Treatment for Military, Police and Veterans
Brief Title: A Trial of an Online Chronic Pain Treatment for Military, Police and Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Jeremiah Buhler, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2016:145
Record Dates: First submitted 2017-09-16; First posted 2017-09-19 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: D059350
Keywords: chronic pain; online treatment; acceptance-based therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Condition (Experimental): An Online 8-week Acceptance-based Behavioural Therapy for chronic pain.
  Interventions: Behavioral: Acceptance-based Behavioural Therapy
- Wait-list Control Condition (No Intervention): Wait-list Control group (8-weeks)

INTERVENTIONS:
Behavioral: Acceptance-based Behavioural Therapy — The treatment program is an eight module (8-week) ABBT for chronic pain. The online treatment material is administered via the WebCAPSI Therapy program. This online program allows participants to progress through the treatment modules at their own pace. Each module is designed to cover a specific component of ABBT and will facilitate understanding of the components through audio files, veteran, military and RCMP-specific vignettes, text-based material, and homework exercises/assignments. Each module is designed to be completed in 60 minutes or less. On the completion of each module, and facilitated through the WebCAPSI Therapy program, the participants are asked to complete a homework exercise to which they answer questions previously encountered throughout the module. The principle therapist responds to each homework exercise within 24-hours of its online submission.
  Arms: Treatment Condition

SUMMARY:
Chronic pain is a serious health issue in Canada. Individuals who experience chronic pain often find it difficult to attend in-person treatment sessions for a variety of reasons including pain flare-ups, discomfort when travelling, pain-induced avoidant behaviours, and time constraints. These factors, if not addressed through appropriate treatment, serve as a detriment to the individual's functioning by maintaining the pain cycle and preventing the individual from engaging in previously enjoyed activities. Online treatments have the potential to assist individuals who would otherwise have difficulty attending in-person treatment sessions. This study evaluated the efficacy of an online acceptance-based behavioural treatment for chronic pain designed for military, police, and veteran populations. Participants (n = 29) were randomized into either a treatment condition or wait-list control condition, and asked to complete a battery of measures which underscore the key facets of the fear-avoidance model of chronic pain. A series of 2 x 2 mixed model ANOVA's revealed statistically significant Time x Condition interactions for pain disability, kinesiophobia, and pain acceptance, as well as statistically significant pre- to post-treatment simple main effect contrasts for pain catastrophizing, kinesiophobia, and pain acceptance. For those in the treatment group, no significant changes in scores were found between post-treatment and three-month follow-up; however, the sample size was too small to draw conclusions regarding this finding. Baseline PTSD and depression scores were found to be significant predictors of change in pain acceptance levels over the course of treatment. Overall, the results support the efficacy of the ABBT treatment for chronic pain for military, police and veterans.

DETAILED DESCRIPTION:
This study is an extension of a pilot study that was conducted investigating an online acceptance-based behavioural therapy (ABBT) for chronic pain. The online treatment runs for a total of 8 weeks and includes interactive content to promote the participant's engagement with the treatment material. The treatment has been specifically tailored for military, police and veteran populations as it uses language and audio vignettes to which military, police and veteran individuals can easily relate. Based on promising results from a pilot study conducted using the online ABBT program, the investigators conducted a randomized control trial (RCT) of the treatment by randomly allocating participants into either a treatment group, or a wait-list control group. Clients who are new to the participating clinic participate in an intake appointment with the clinic's intake nurse, and during this appointment are informed about the different research projects currently being run at the clinic. Participants interested in the study were screened for inclusion and exclusion criteria during their intake appointment. For this study, all eligible participants were asked to complete an informed consent form prior to being issued a unique password and user ID for access to the online portion of the treatment. A treatment fidelity plan and data safety monitoring plan have been established to ensure treatment procedures remain consistent across groups, and that data integrity is monitored over the duration of the study. The treatment program is an eight module (8-week) ABBT for chronic pain. The online treatment material is administered via the WebCAPSI Therapy program. This is an online password-protected program which allows participants to progress through the treatment modules at their own pace. Each module is designed to cover a specific component of ABBT and facilitated understanding of the components through audio files, veteran, military and RCMP-specific vignettes, text-based material, and homework exercises/assignments. Each module is designed to be completed in 60 minutes or less and participants have the option to return to the program and the modules as often as they like during the course of the treatment period. On the completion of each module, and facilitated through the WebCAPSI Therapy program, the participants are asked to complete a homework exercise to which they answer questions previously encountered throughout the module. The principle therapist responds to each homework exercise within 24-hours of its online submission, with feedback and encouragement. The participants completed a battery of measures at the outset of the randomization process (both treatment and wait-list control conditions), and again at the end of the 8-weeks. A 3-month follow-up assessment was conducted to evaluate the maintenance of treatment gains. Only participants who complete at least 5 out of the 8 modules were considered to have "completed" the treatment, and therefore included in the analyses. The interactions from the mixed model ANOVA analyses were statistically significant for changes in pain interference, kinesiophobia, and pain acceptance. Regarding the main effects of Time, only change in pain acceptance was found to be significant, whereas no main effect of Condition was found to be statistically significant. For the treatment condition, dependent t-tests were conducted to further assess mean differences between the pre-treatment, post-treatment, and follow-up scores on each of the four dependent variables. The results for the pre- to-post-test dependent t-tests revealed statistically significant differences for all of the dependent variables except for pain interference, although even this measurement was close to statistical significance with t(13) = 2.07, p = .059. As expected, there were no statistically significant differences between post-treatment and follow-up for each of the dependent variables. Only change in pain acceptance scores was significantly predicted by participants scores on both measures of PTSD and depression symptoms. The results from this study provide further empirical support for the use of acceptance-based behavioural interventions for treating various chronic pain conditions, and thus add to the recent growing body of literature for acceptance-based treatments for chronic pain. These results also highlight how this acceptance-based behavioural treatment helps to significantly decrease pain interference and kinesiophobia, as well as increase pain acceptance. This study adds a unique contribution to the understanding of how depression and PTSD symptoms influence treatment gains for pain acceptance, when utilizing an acceptance-based behavioural intervention for chronic pain. These positive findings provide further support for the use of this acceptance-based behavioural treatment for chronic pain within police and military populations.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be individuals who have reported chronic pain lasting longer than 6 months, and who have been referred for treatment at the OSIC. Participants, male or female, will be either an active RCMP officer, an active member of the Canadian Forces, or a veteran of the Canadian Forces or RCMP. The participants will be required to have access to a computer with internet access for a minimum of 60 minutes per week.

Exclusion Criteria:

* Any individual who does not meet the requirements listed above is not eligible for this study. Likewise, any individual with seriously impaired concentration, psychosis, suicidality, unstable living situation, or any other similar disorder or condition that would render them unfit for a self-help based treatment will not be considered eligible for this study. Potential participants who neither read nor write in English, as well as those who are unable to provide informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Pain Disability Index | 8 weeks
  The Pain Disability Index (PDI) is a 7-item scale which captures the respondent's perceived interference pain plays in their lives in 7 domains: family/home responsibilities recreation, social activity, occupation, sexual behavior, self-care, and life-support activity.
Chronic Pain Acceptance Questionnaire | 8 weeks
  The Chronic Pain Acceptance Questionnaire (CPAQ), a 20-item scale designed to measure acceptance in individuals dealing with pain.
The Pain Catastrophizing Scale | 8 weeks
  The Pain Catastrophizing Scale (PCS) is a short 13-item measure which evaluates the pain-related catastrophizing behaviours and cognitions of individuals.
The Tampa Scale for Kinesiophobia | 8 weeks
  The Tampa Scale for Kinesiophobia (TSK-11) 11-item version is a self-report measure that contains 11 questions designed to assess a client's fear of movement and re-injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Operational Stress Injury Clinic, Winnipeg, Manitoba, Canada